CLINICAL TRIAL: NCT07207291
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of JKN2501 for Injection in Chinese Healthy Volunteers
Brief Title: Phase I Study of Single/Multiple Ascending Doses of JKN2501 for Injection in Chinese Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Joincare Pharmaceutical Group Industry Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JKN2501-I-01
Record Dates: First submitted 2025-09-04; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Bacterial Infections; Urinary Tract Infections; Intra-Abdominal Infections; Respiratory Tract Infections
Keywords: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections; Urinary Tract Infections; Intraabdominal Infections; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SAD Cohort1 (Experimental): JKN2501 125mg only, without placebo.
  Interventions: Drug: JKN2501
- SAD Cohort2 (Experimental): JKN2501 B mg
  Interventions: Drug: JKN2501; Drug: Placebo
- SAD Cohort3 (Experimental): JKN2501 C mg
  Interventions: Drug: JKN2501; Drug: Placebo
- SAD Cohort4 (Experimental): JKN2501 D mg
  Interventions: Drug: JKN2501; Drug: Placebo
- SAD Cohort5 (Experimental): JKN2501 E mg
  Interventions: Drug: JKN2501; Drug: Placebo
- MAD Cohort1 (Experimental): JKN2501 F mg
  Interventions: Drug: JKN2501; Drug: Placebo
- MAD Cohort2 (Experimental): JKN2501 G mg
  Interventions: Drug: JKN2501; Drug: Placebo
- MAD Cohort3 (Experimental): JKN2501 H mg
  Interventions: Drug: JKN2501; Drug: Placebo

INTERVENTIONS:
Drug: JKN2501 — Administration: Intravenous (IV) infusion.
Drug: Placebo — 0.9% Sodium Chloride Injection as Placebo. Administration: Intravenous (IV) infusion.
  Arms: MAD Cohort1; MAD Cohort2; MAD Cohort3; SAD Cohort2; SAD Cohort3; SAD Cohort4; SAD Cohort5

SUMMARY:
This Phase I study is a randomized, double-blind, placebo-controlled, dose-escalation trial conducted at a single center. It consists of two parts:

Part 1 (SAD): Evaluates the safety, tolerability, and pharmacokinetics (PK) of single ascending intravenous doses of JKN2501 in healthy adults. Biological samples (blood, urine, feces) will be collected for PK analysis.

Part 2 (MAD): Evaluates the safety, tolerability, and PK of multiple ascending intravenous doses of JKN2501 in healthy adults.

Dose levels may be adjusted based on emerging safety, tolerability, and PK data from preceding cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent; able to comply with study requirements and communicate effectively.
* Healthy subjects aged 18-45 years (inclusive) at screening.
* BMI 19.0-26.0 kg/m² (inclusive); weight ≥50 kg (male) or ≥45 kg (female).
* Vital signs, physical examination, ECG, laboratory tests, chest X-ray, and abdominal ultrasound results judged as normal or clinically insignificant by the investigator.
* Agreement to use effective non-pharmaceutical contraception from signing ICF until 90 days after last dose; no sperm/egg donation plans during this period.

Exclusion Criteria:

* Pregnant/lactating women; positive pregnancy test; unprotected sex within 2 weeks prior to dosing.
* Investigator-determined history or presence of clinically significant disorder that may affect safety or trial participation.
* Use of drugs known to inhibit/induce hepatic metabolism within 4 weeks, or any medication (prescription, OTC, herbal, vitamins) within 2 weeks prior to dosing; planned use during the trial.
* Major surgery within 3 months prior to screening or planned during trial; history of surgery potentially affecting results.
* History of febrile illness or active infection within 2 weeks prior to screening.
* Blood loss/donation >400 mL within 3 months prior to screening, or received blood products; plans to donate blood during trial or within 30 days after last dose.
* History of significant food/drug allergy, or allergy to JKN2501/excipients.
* Excessive alcohol consumption; inability to abstain from alcohol from 48h pre-dose until end of study.
* Smoking ≥5 cigarettes/day within 3 months prior to screening; inability to abstain from smoking from 48h pre-dose until end of study.
* History of drug abuse; positive urine drug screen at baseline (Day -1).
* Positive alcohol breath test at baseline (Day -1).
* Participation in another interventional clinical trial within 3 months prior to screening or planned during this trial.
* Estimated glomerular filtration rate (eGFR) <90 mL/min.
* Serum total calcium below lower limit of normal at screening.
* Investigator-determined unsuitable venous access for PK sampling/infusion, or history of adverse symptoms/phobias related to infusion/phlebotomy.
* Excessive daily intake of tea, coffee, or caffeinated beverages within 3 months prior to screening.
* Consumption of grapefruit, Seville oranges, caffeine, or xanthine-rich foods/beverages within 48h prior to first dose; inability to abstain during the trial.
* History of QTc prolongation; or investigator-determined clinically significant ECG abnormalities at screening/baseline.
* Any other condition deemed by the investigator to make the subject unsuitable for participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple intravenous (IV) infusions of JKN2501 for Injection in healthy adults. | SAD: Baseline to Day 8 post-dose. MAD: Baseline to Day 18 post-dose.
  Number of participants with treatment-related adverse events as assessed by CTCAE V5.0.
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.

SECONDARY OUTCOMES:
Pharmacokinetic parameter of JKN2501: Tmax | SAD: Baseline to Day 8 post-dose. MAD: Baseline to Day 18 post-dose.
Pharmacokinetic parameter of JKN2501: Cmax | SAD: Baseline to Day 8 post-dose. MAD: Baseline to Day 18 post-dose.
Pharmacokinetic parameter of JKN2501: t1/2 | SAD: Baseline to Day 8 post-dose. MAD: Baseline to Day 18 post-dose.
Pharmacokinetic parameter of JKN2501: AUC0-t | SAD: Baseline to Day 8 post-dose. MAD: Baseline to Day 18 post-dose.
Pharmacokinetic parameter of JKN2501: AUC0-∞ | SAD: Baseline to Day 8 post-dose. MAD: Baseline to Day 18 post-dose.
Pharmacokinetic parameter of JKN2501: CL | SAD: Baseline to Day 8 post-dose. MAD: Baseline to Day 18 post-dose.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No